CLINICAL TRIAL: NCT03452917
Title: Randomized Clinical Trial of Sodium Nitrite for Out of Hospital Cardiac Arrest
Brief Title: Clinical Trial of Sodium Nitrite for Out of Hospital Cardiac Arrest
Acronym: SNOCAT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Francis Kim, Professor, Medicine/Division of Cardiology, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 51605; R01HL129722 (NIH)
Record Dates: First submitted 2018-02-12; First posted 2018-03-02 (Actual); Results first posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-04

CONDITIONS: Out-Of-Hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest | interventions — Sodium Nitrite

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 2 ml of normal saline (n=500)
  Interventions: Drug: Placebo
- sodium nitrite (Experimental): 45 mg IV of sodium nitrite (n=500) or 60 mg IV sodium nitrite (n=500) given during active resuscitation from out of hospital cardiac arrest.
  Interventions: Drug: sodium nitrite 45 mg; Drug: sodium nitrite 60 mg

INTERVENTIONS:
Drug: Placebo — 500 patients will 2 ml of normal saline
  Arms: Placebo
Drug: sodium nitrite 45 mg — 500 patients will receive 45 mg IV sodium nitrite
  Arms: sodium nitrite
Drug: sodium nitrite 60 mg — 500 patients will receive a dose of 60 mg IV sodium nitrite
  Arms: sodium nitrite

SUMMARY:
In this clinical study, a total of 1500 patients with out-of-hospital cardiac arrest in Seattle/King County will be enrolled. This will be a randomized clinical trial and patients will receive either two different doses of IV sodium nitrite (45 mg or 60 mg) or placebo during resuscitation in the field by paramedics. The primary outcome will be proportion of patients surviving to hospital admission.

DETAILED DESCRIPTION:
The hemodynamic effects of the optimal dose of IV nitrite administered in patients with cardiac arrest are unknown. A significant negative hemodynamic effect from nitrite would decrease the proportion of patients admitted to the hospital, increase rate of re-arrest, or increase the need for vasopressor support in the field. In Seattle/King County, typically 40% of out-of-hospital cardiac arrest patients attended to by paramedics have Return of spontaneous circulation (ROSC) and are admitted to the hospital. In this study, 1500 patients with out-of-hospital cardiac arrest who are undergoing resuscitation by paramedics will be randomized to receive placebo (n=500) or 45 mg IV (n=500) or 60 mg dose (n=500) of sodium nitrite. The study will have 80% power to detect an absolute increase in hospital admission rate of 8% (1-sided .05 level test for each of the two comparisons (45 mg vs placebo and 60 mg vs placebo, no adjustment for multiple comparisons), with a hospital admission rate of 40% in the placebo group and with one interim analysis and stopping only for potential futility and/or harm). The investigators will examine the proportion of patients who survive to discharge as a secondary measure of efficacy.

Patients will be eligible for this study if:

1. Intravenous access (IV)/intraosseous access(IO)
2. Cardiac arrest, either Ventricular Fibrillation (VF) or non-VF patients receiving Advanced Cardiac Life Support (ACLS) by Seattle/King County paramedics.
3. Age 18 years or older
4. Comatose

Exclusion Criteria

1. Traumatic cause of cardiac arrest
2. Prisoner, pregnancy, age less than 18 (special population/vulnerable population)
3. Known DNAR
4. Drowning as cause of arrest.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac arrest, either VF or non-VF, patients receiving ACLS by paramedics
* IV or IO access
* Comatose

Exclusion Criteria:

* traumatic cause of cardiac arrest
* prisoner, pregnancy
* known DNAR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1502 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis Kim, MD, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim F, Maynard C, Dezfulian C, Sayre M, Kudenchuk P, Rea T, Sampson D, Olsufka M, May S, Nichol G. Effect of Out-of-Hospital Sodium Nitrite on Survival to Hospital Admission After Cardiac Arrest: A Randomized Clinical Trial. JAMA. 2021 Jan 12;325(2):138-145. doi: 10.1001/jama.2020.24326. PMID 33433575

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1502 were enrolled. A total of 1497 were randomized. 5 patients were excluded due to missing kit information.
Groups:
- Sodium Nitrite 45 mg: 45 mg IV of sodium nitrite (n=500)
- Sodium Nitrite 60 mg: sodium nitrite 60 mg (n=500)
Period: Overall Study
Arm/Group | Placebo | Sodium Nitrite 45 mg | Sodium Nitrite 60 mg
Started | 499 | 500 | 498
Completed | 499 | 500 | 498
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 5 patients were excluded since they were incarcerated or were less than 18 years of age. We were not allowed to use their data. There were 1492 patients available for analysis.
Groups:
- Placebo: 2 ml of normal saline
  Placebo: 500 patients will 2 ml of normal saline
- Sodium Nitrite 45 mg: 45 mg IV of sodium nitrite
- Sodium Nitrite 60 mg: 60 mg IV sodium nitrite
- Total: Total of all reporting groups
Arm/Group | Placebo | Sodium Nitrite 45 mg | Sodium Nitrite 60 mg | Total
Number analyzed (Participants) | 496 | 499 | 497 | 1492
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 0 | 1
  Between 18 and 65 years | 222 | 242 | 254 | 718
  >=65 years | 274 | 256 | 243 | 773
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 67 [55 to 76] | 65 [56 to 76] | 64 [52 to 76] | 65 [55 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 165 | 170 | 167 | 502
  Male | 331 | 329 | 330 | 990
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 14 | 10 | 36
  Not Hispanic or Latino | 186 | 201 | 192 | 579
  Unknown or Not Reported | 298 | 284 | 295 | 877
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 271 | 288 | 273 | 832
  Black | 49 | 58 | 51 | 158
  Asian | 38 | 39 | 31 | 108
  Other | 3 | 5 | 2 | 10
  Unknown | 135 | 109 | 140 | 384
Region of Enrollment [Number; unit: participants]
  United States | 496 | 499 | 497 | 1492

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Survived to Hospital Admission
Description: Patient has sustained pulse at arrival to the emergency department
Time Frame: within 24 hours after out of hospital cardiac arrest
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Sodium Nitrite 45 mg | Sodium Nitrite 60 mg
Number analyzed (Participants) | 496 | 499 | 497
Participants | 218 | 205 | 212
Statistical Analysis 1: Comparison: Placebo vs Sodium Nitrite 45 mg; Test type: Superiority; p = 0.82, Chi-squared; Mean Difference (Final Values) = -2.9, 95% CI 1-sided [lower limit -8.0]
Statistical Analysis 2: Comparison: Placebo vs Sodium Nitrite 60 mg; Test type: Superiority; p = 0.66, Chi-squared; Mean Difference (Final Values) = -1.3, 95% CI 1-sided [lower limit -6.5]

2. Secondary Outcome: Survival to Discharge
Description: Patient alive at time of discharge from hospital
Time Frame: within 3-6 months after cardiac arrest
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Sodium Nitrite 45 mg | Sodium Nitrite 60 mg
Number analyzed (Participants) | 496 | 499 | 497
Participants | 74 | 66 | 72
Statistical Analysis 1: Comparison: Placebo vs Sodium Nitrite 45 mg; Test type: Superiority; p = 0.44, Chi-squared; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-6.0 to 2.6]
Statistical Analysis 2: Comparison: Placebo vs Sodium Nitrite 60 mg; Test type: Superiority; p = 0.85, Chi-squared; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-4.9 to 4.0]

3. Secondary Outcome: Number of Days in ICU
Description: Number of days the patient is admitted to the Intensive Care Unit
Time Frame: Within first 3 months of hospital admission
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Sodium Nitrite 45 mg | Sodium Nitrite 60 mg
Number analyzed (Participants) | 496 | 499 | 497
days | 6.7 (8.1) | 8.9 (10.4) | 7.3 (7.2)
Statistical Analysis 1: Comparison: Placebo vs Sodium Nitrite 45 mg; Test type: Superiority; p = 0.12, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 2.2, 95% CI 2-sided [-0.9 to 5.4]
Statistical Analysis 2: Comparison: Placebo vs Sodium Nitrite 60 mg; Test type: Superiority; p = 0.41, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-2.5 to 3.6]

4. Secondary Outcome: Survival to 24 Hours
Description: Patient is alive after the first 24 hours after admission to the hospital
Time Frame: within first 24 h after hospital admission
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Sodium Nitrite 45 mg | Sodium Nitrite 60 mg
Number analyzed (Participants) | 496 | 499 | 497
Participants | 181 | 170 | 171
Statistical Analysis 1: Comparison: Placebo vs Sodium Nitrite 45 mg; Test type: Superiority; p = 0.42, Chi-squared; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-8.3 to 3.5]
Statistical Analysis 2: Comparison: Placebo vs Sodium Nitrite 60 mg; Test type: Superiority; p = 0.49, Chi-squared; Mean Difference (Final Values) = -2.1, 95% CI 2-sided [-8.0 to 3.9]

5. Secondary Outcome: Re-arrest
Description: Patient loses pulses during transport to the hospital. Event occurs before admission to hospital.
Time Frame: before hospital arrival
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Sodium Nitrite 45 mg | Sodium Nitrite 60 mg
Number analyzed (Participants) | 291 | 270 | 294
Participants | 139 | 130 | 156
Statistical Analysis 1: Comparison: Placebo vs Sodium Nitrite 45 mg; Test type: Superiority; p = 0.93, Chi-squared; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-7.8 to 8.6]
Statistical Analysis 2: Comparison: Placebo vs Sodium Nitrite 60 mg; Test type: Superiority; p = 0.20, Chi-squared; Mean Difference (Final Values) = 5.3, 95% CI 2-sided [-2.8 to 13.3]

6. Secondary Outcome: Survival to 48 Hours After Admission to Hospital
Description: Patient is alive after first 48 hours after admission to the hospital
Time Frame: within first 48 hours after admission to hospital
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Sodium Nitrite 45 mg | Sodium Nitrite 60 mg
Number analyzed (Participants) | 496 | 499 | 497
Participants | 161 | 152 | 151
Statistical Analysis 1: Comparison: Placebo vs Sodium Nitrite 45 mg; Test type: Superiority; p = 0.50, Chi-squared; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-7.7 to 3.8]
Statistical Analysis 2: Comparison: Placebo vs Sodium Nitrite 60 mg; Test type: Superiority; p = 0.48, Chi-squared; Mean Difference (Final Values) = -2.1, 95% CI 2-sided [-7.8 to 3.7]

7. Secondary Outcome: Survival to 72 Hours After Admission to Hospital
Description: Patient is alive after first 72 hours after admission to the hospital
Time Frame: within first 72 hours after admission to hospital
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Sodium Nitrite 45 mg | Sodium Nitrite 60 mg
Number analyzed (Participants) | 496 | 499 | 497
Participants | 142 | 133 | 131
Statistical Analysis 1: Comparison: Placebo vs Sodium Nitrite 45 mg; Test type: Superiority; p = 0.49, Chi-squared; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-6.0 to 2.6]
Statistical Analysis 2: Comparison: Placebo; Test type: Superiority; p = 0.85, Chi-squared; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-4.9 to 4.0]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time period of randomization to hospital discharge
Description: Other variables (rate of rearrest, use of norepinephrine in the filed) were chosen as respecified safety outcomes
  There were no unexpected adverse events observed in this study. Of note, this is not atypical for studies of out of hospital cardiac arrest, because it is very difficult to identify and observe adverse events for patients whose heart has stopped beating.
Arm/Group | Placebo | Sodium Nitrite 45 mg | Sodium Nitrite 60 mg
All-Cause Mortality (participants affected / at risk) | 422/496 | 433/499 | 425/497
Serious Adverse Events (participants affected / at risk) | 280/496 | 249/499 | 268/497
Other Adverse Events (participants affected / at risk) | 21/496 | 19/499 | 15/497
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=496) | Sodium Nitrite 45 mg (N=499) | Sodium Nitrite 60 mg (N=497)
Re-arrest first 24 hours of hospitalization (Cardiac disorders) | 76 (76) | 65 (65) | 74 (74) — Loss of pulse during hospitalization. Includes all patients, including patients who died before emergency room or hospitalization.
Pressors in first 24 hours after hospitalization (Cardiac disorders) | 190 (190) | 173 (173) | 185 (185) — Use of any pressors to support blood pressure during first 24 hours. The denominator includes patients who died in the emergency department or before admission to the hospital
sustained hypotension in hospital, first 24 hours (Cardiac disorders) | 14 (14) | 11 (11) | 9 (9) — Systolic blood pressure of less than 90 mmHg during first 24 hours after randomization.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=496) | Sodium Nitrite 45 mg (N=499) | Sodium Nitrite 60 mg (N=497)
Positive troponin (Cardiac disorders) | 21 (21) | 19 (19) | 15 (15) — Troponin level greater than 0.02-0.08 ng/ml at any time during hospitalization Post hoc safety measure The denominator includes patients who died in the emergency department or died before admission to the hospital.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-31): https://cdn.clinicaltrials.gov/large-docs/17/NCT03452917/Prot_SAP_000.pdf